CLINICAL TRIAL: NCT03307460
Title: Phase II Trial: uPAR-PET/MR in Patients With Newly Diagnosed Prostate Cancer; Non-invasive Characterization of Tumor Aggressiveness
Brief Title: uPAR-PET/MRI in Patients With Prostate Cancer for Evaluation of Tumor Aggressiveness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marie Øbro Fosbøl, Medical doctor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK-2017-PC-1; 2017-002276-37 (EudraCT Number)
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uPAR PET/MRI (Experimental): 68Ga-NOTA-AE105 is injected once for performing a PET/MRI scan
  Interventions: Drug: 68Ga-NOTA-AE105

INTERVENTIONS:
Drug: 68Ga-NOTA-AE105 — PET/MRI scan
  Other Names: PET/MRI

SUMMARY:
Prospective study to evaluate the value of uPAR-targeted PET/MR scan using the tracer 68Ga-NOTA-AE105 in patients with newly diagnosed prostate cancer

DETAILED DESCRIPTION:
Prostate cancer is one of the most frequent types of cancer in men. The characteristics of the disease varies significantly among patients where some have an indolent type of cancer, from which they will never experience symptoms while others have highly aggressive malignant disease that requires prompt therapeutic action.

Treatment of localized prostate cancer is based on a risk stratification, where patients are either offered therapy with curative intent - surgery or radiotherapy - or in case of low-risk disease an "active surveillance" strategy can be advised. In active surveillance the disease is monitored by PSA measurement, repeated biopsies and digital rectal examination. Some patients progress during active surveillance to a higher risk classification, which may lead to selection of active therapy.

The aim of this study is to investigate positron emission tomography (PET) with the radiolabelled tracer 68Ga-NOTA-AE105, combined with magnetic resonance imaging (MRI) in patients with newly diagnosed prostate cancer. 68Ga-NOTA-AE105 targets the receptor urokinase-type plasminogen activator receptor (uPAR), which is a known marker for aggressive disease in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified prostate cancer
* Capable of understanding written information and giving informed consent
* Planned to enter active surveillance strategy or undergo therapy with curative intent (surgery or radiotherapy)

Exclusion Criteria:

* Obesity (Body weight over 140 kg)
* Known allergy to 68-Ga-NOTA-AE105
* Metallic components in the body that contradicts MRI scan
* Severe claustrophobia making the person unable to complete an MRI scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlation with Gleason Score | 3 months after PET/MRI
  Correlate the uptake of 68Ga-NOTA-AE105 with Gleason Score obtained from biopsy material.

SECONDARY OUTCOMES:
Prognostic value | 3 years from PET/MRI
  Evaluate the prognostic value of uPAR PET/MRI in patients with prostate cancer either undergoing therapy with curative intent or active surveillance.
Diagnostic accuracy in staging lymph nodes | 3 months from PET/MRI
  Evaluate the diagnostic accuracy of uPAR PET/MRI in identifying regional lymph node metastases in patients with newly diagnosed prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ø Fosboel, MD, Principal Investigator — Rigshospitalet, Department of Clinical Physiology, Nuclear Medicine & PET
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided